CLINICAL TRIAL: NCT04257812
Title: Monitoring of Ceftolozane-Tazobactam Plasmatic Levels in Critical Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Other Study IDs: FIS-CEF-2019-01
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-01

CONDITIONS: Serious Infection
Keywords: Ceftolozane-Tazobactam; Plasmatic Levels; Serious Infection; Dose adjustment
MeSH Terms: interventions — ceftolozane, tazobactam drug combination

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ceftolozane-Tazobactam cohort: Patients older than 18 years old that are hospitalised in the Virgen Macarena University Hospital that are being treated with Ceftolozane-Tazobactam in empiric or targeted treatment.
  Interventions: Drug: Ceftolozane/tazobactam

INTERVENTIONS:
Drug: Ceftolozane/tazobactam — The dose will be 1g ceftolozane + 0,5 g tazobactam every 8 hours or 2 g ceftolozane + 1 g tazobactam, it´s recommended to use this last dose regimen in patients with pneumonia or septic shock of any focus.
  The patients will be followed as it´s done habitually. There will be done infection focus cultures and others according to usual clinical practice. It´ll be determined the clinical response and mortality in the days 14 and 30 after the beginning of the medicine, respectively.
  The Ceftolozane-Tazobactam levels determination will always be made in state of equilibrium (after the third dose). Four samples will be collected:
  1. Just before the antibiotic infusion.
  2. One hour after the antibiotic infusion.
  3. Three hours after the antibiotic infusion.
  4. Six hours after the antibiotic infusion.

SUMMARY:
The aim of this study is to determine the Ceftolozane-Tazobactam Plasmatic Levels and and analyse the clinical impact that might have the dose regimens that have been used until now.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old.
* Hospitalised for a serious illness.
* Treated with Ceftolozane-Tazobactam
* Patients that signed the Informed Consent.

Exclusion Criteria:

* Allergic to any component of Ceftolozane-Tazobactam.
* Any surgical or medical evidence that according to the investigator could interfere with the pharmacodynamics of the medication: absorption, distribution, metabolism or excretion.
* Concomitant terminal illness.
* Unable to sign the Informed Consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years old, hospitalised in the Virgen Macarena University Hospital for a serious infection that meet all the inclusion criteria and none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-02-15 (Estimated); Primary Completion 2021-03-15 (Estimated); Study Completion 2022-06-15 (Estimated)

PRIMARY OUTCOMES:
Determine the Ceftolozane-Tazobactam seric concentrations and analyse the clinic impact that could have the dose regimens used until now. | Up to 12 months after the antibiotic administration
  Determination of the Ceftolozane-Tazobactam seric concentration by collecting 4 blood samples and measuring its antibiotic levels and if it´s achieved an adequate therapeutic efficacy assessed by the patient´s clinical and microbiological recovery.
  The dose regimens used until now are 1+0,5 g every 8 hours in case of intra-abdominal infection or complicated urinary infection and 2 +1 g every 8 hours in case of pneumonia or septic shock of any focus.

SECONDARY OUTCOMES:
Analyse if with both dose regimens are achieved the PK/PD parameters associated with the maximum therapeutic efficacy in patients with renal hyper clearance. | Up to 12 months after the antibiotic administration
  Determine if with both dose regimens are achieve the pharmacodynamic and pharmacokinetic parameters associated with the maximum therapeutic efficacy in patients that have creatinine clearance above 130 ml/min.
Determine the Ceftolozane-Tazobactam seric concentrations and analyse if with both dose regimens are achieved the PK/PD parameters associated with the maximum therapeutic efficacy in patients with morbid obesity. | Up to 12 months after the antibiotic administration
  Determination of the Ceftolozane-Tazobactam seric concentration by collecting 4 blood samples and measuring its antibiotic levels and if with both dose regimens are achieve the pharmacodynamic and pharmacokinetic parameters associated with the maximum therapeutic efficacy in patients that have BMI (body mass index) above 40
Determine the Ceftolozane-Tazobactam seric concentrations and analyse if with both dose regimens are achieved the PK/PD parameters associated with the maximum therapeutic efficacy in patients with continuous renal replacement technique. | Up to 12 months after the antibiotic administration
  Determination of the Ceftolozane-Tazobactam seric concentration by collecting 4 blood samples and measuring its antibiotic levels and if with both dose regimens are achieve the pharmacodynamic and pharmacokinetic parameters associated with the maximum therapeutic efficacy in patients that have their blood purified extracorporeally, replacing the renal function continuously 24 hours of the day.
Determine if in patients with Gram-negative bacillary bacteremia are achieved concentrations that are 100 % of the time 4 times above the minimum inhibitory concentration (MIC). | Up to 12 months after the antibiotic administration
  Determination of if in patients with Gram-negative bacillary bacteremia (patients with their bloodstream invaded by Gram-negative bacillary which is diagnosed by blood culture) are achieved concentrations that are 100 % of the time 4 times above the MIC by strips of isolated pathogen gradient .
Determine by a Monte Carlo simulation model the dose regimen that should be used. | Up to 12 months after the antibiotic administration
  Determination by a Monte Carlo simulation model of the dose regimen that should be used based on the pharmacokinetic parameters and according to the defined efficacy pharmacodynamic parameters.
Describe the frequency of resistance´s development during the Ceftolozane-Tazobactam treatment and, if it´s possible to evaluate if there´s a correlation with the seric levels. | Up to 12 months after the antibiotic administration
  Description of the rate of resistance´s development during the Ceftolozane-Tazobactam and if there´s a correlation with the Ceftolozane-Tazobactam seric levels.
Describe the Ceftolozane-Tazobactam treatment´s clinical result as well as existence of adverse effects. | Up to 12 months after the antibiotic administration
  Description of the Ceftolozane-Tazobactam clinical results as well as the rate and seriousness of adverse effects.

CONTACTS AND LOCATIONS:
Overall Officials: José Garnacho Montero, Principal Investigator — Hospital Universitario Virgen Macarena
Locations (1):
- Hospital Universitario Virgen Macarena, Seville, Spain